CLINICAL TRIAL: NCT05604209
Title: IGHID 12107 - A Phase I Study to Evaluate the Safety and Immunogenicity of the ChAdOx1.HIVconsv62 - MVA.tHIVconsv4 (C62-M4) or, ChAdOx1.tHIVconsv1+C62 - MVA.tHIVconsv3+M4 (C1C62-M3M4) Prime-Boost Regimens in Persons With HIV-1 Suppressed on Antiretroviral Therapy
Brief Title: Safety and Immunogenicity of HIV-1 Vaccines C62-M4 or C1C62-M3M4 in Persons With HIV-1 Suppressed on ART
Acronym: CM HIV-CORE008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0094; 5U01AI131310 (NIH); IGHID 12107 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2022-10-27; First posted 2022-11-03 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-04

CONDITIONS: HIV Vaccine; HIV-1-infection
Keywords: Vaccination; Immunogenicity; HIV-1; HIV vaccine; HIV; MVA; ChAdOx1; T-cell vaccine; Therapeutic T-cell vaccine
MeSH Terms: interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 8:8:2 to one of three study arms (C62-M4, C1C62-M3M4, Placebo) and receive study treatment or placebo at Days 0 and 28.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- C62-M4 (Experimental): ChAdOx1.HIVconsv62 (C62) vaccine administered at Day 0, followed by MVA.tHIVconsv4 (M4) vaccine administered at Day 28
  Interventions: Biological: ChAdOx1.HIVconsv62; Biological: MVA.tHIVconsv4
- C1C62-M3M4 (Experimental): ChAdOx1.tHIVconsv1 (C1) and ChAdOx1.HIVconsv62 (C62) vaccines administered at Day 0, followed by MVA.tHIVconsv3 (M3) and MVA.tHIVconsv4 (M4) vaccines administered at Day 28
  Interventions: Biological: ChAdOx1.HIVconsv62; Biological: ChAdOx1.tHIVconsv1; Biological: MVA.tHIVconsv4; Biological: MVA.tHIVconsv3
- Placebo (Placebo Comparator): Placebo administered on Day 0 and Day 28
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ChAdOx1.HIVconsv62 — Administered intramuscularly (IM) at Day 0
  Arms: C1C62-M3M4; C62-M4
Biological: ChAdOx1.tHIVconsv1 — Administered intramuscularly (IM) at Day 0
  Arms: C1C62-M3M4
Biological: MVA.tHIVconsv4 — Administered intramuscularly (IM) at Day 28
  Arms: C1C62-M3M4; C62-M4
Biological: MVA.tHIVconsv3 — Administered intramuscularly (IM) at Day 28
  Arms: C1C62-M3M4
Other: Placebo — Administered at intramuscularly (IM) Day 0 and Day 28
  Other Names: Normal saline; Sodium chloride
  Arms: Placebo

SUMMARY:
This is a double blind, randomized, placebo-controlled, parallel design study in which 18 in participants with HIV (PWH) on suppressive antiretroviral therapy will be randomly assigned to receive vaccination with C62 followed by M4 (C62-M4), C62 and C1 followed by M4 and M3 (C1C62-M3M4), or placebo.

The purpose of this study is to find out:

* If it is safe for people to receive intramuscular (IM) vaccination with C62-M4 or C1C62-M3M4
* If giving participants these vaccine doses will improve their immune system response to help the body get rid of HIV in the cells

DETAILED DESCRIPTION:
This is a Phase 1, double blind, randomized to evaluate safety and immunogenicity of investigational vaccines given in a sequential regimen.

Participants will be screened for eligibility and have a enrollment visit with leukapheresis (white blood cell collection procedure). After determination of eligibility, participants will be randomized on Day 0 to C62-M4, C1C62-M3M4, or placebo arms in a 8:8:2 ratio. C62, C1C62, or placebo will be given as an intramuscular (IM) injection on Day 0. M4, M3M4, or placebo will be given as an IM injection on Day 28. Post-treatment leukapheresis will be completed at Day 56.

Each enrolled participant will complete 12 clinic study visits and 5 phone study visits over the course of approximately 36 weeks (9 months).

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral assay.

   A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

   Note: The term "licensed" refers to a US FDA-approved kit, which is required for all IND studies. World Health Organization (WHO) and Centers for Disease Control and Prevention (CDC) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment.
2. Ages = 18 to = 70 years old
3. Able and willing to give written informed consent.
4. Able and willing to provide adequate locator information.
5. Able and willing to comply with all study requirements through D196 Week 28.
6. Continuous antiretroviral therapy (ART) prior to screening, defined as not missing more than 14 total days and never more than 7 consecutive days in the last 3 months prior to screening.
7. No change in any ART medication in the 30 days prior to screening.

   Permitted ART regimens include:
   1. At least 3 ART agents (not counting ritonavir or cobicistat as one of the agents if less than a 200 mg total daily dose). One of the agents must include an integrase inhibitor, NNRTI (Non-Nucleoside Reverse Transcriptase Inhibitors), or a boosted-PI (protease inhibitor).

      OR
   2. Two (2) ART agents in which one of the agents is either a boosted protease inhibitor or an integrase inhibitor.

   Note: Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis. Note: Changes in drug formulation or dose are allowed (e g, tenofovir disoproxil fumarate (TDF) to tenofovir alafenamide (TAF), ritonavir to cobicistat or separate ART agent dosing to fixed-dose combination), but none within 30 days prior to screening.

   Note: Prior changes in, or elimination of, medications for easier dosing schedule, intolerance, toxicity, an improved side effect profile or within a drug class are permitted if an alternative suppressive regimen was maintained, but not within 30 days prior to screening.
8. Ability and willingness of participant to continue ART throughout the study.
9. Plasma HIV-1 RNA <50 copies/mL at 2 time points in the 24 months prior to screening and never =50 copies/mL on 2 consecutive time points in the last 24 months.

   Note: Plasma HIV-1 RNA must be performed by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
10. Documented plasma HIV-1 RNA result <50 copies/mL =24 months but = 36 months prior to screening.
11. Plasma HIV-1 RNA level <50 copies/mL on an FDA-approved HIV RNA assay performed at a US CLIA Certified Laboratory (or its equivalent) at screening.
12. CD4 cell count = 350 cells/mm3 performed at any US laboratory that has a CLIA certification or its equivalent at screening.
13. Completion of COVID-19 vaccine dosing at least 14 days prior to enrollment (see exclusion criterion regarding COVID-19 vaccination).
14. Hepatitis C (HCV) antibody negative result at screening or, if the participant is HCV antibody positive, a negative HCV RNA at screening.
15. Hepatitis B surface antigen (HBsAg) negative at screening.
16. Adequate vascular access for leukapheresis.
17. Able and willing to receive IM injections in both arms without difficulty.
18. All women must have a negative serum pregnancy test with a sensitivity of a least 25 U/mL at screening regardless of reproductive potential.
19. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) while on study.

    Note: Women of child-bearing potential is defined as women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy
20. All men and women participating in sexual activity that could lead to pregnancy must agree to consistently use at least one of the following forms of birth control for at least 21 days prior to Visit 4 (D0) and for 4 months after their last vaccination:

    1. Condoms (male or female) with or without a spermicidal agent
    2. Diaphragm or cervical cap with spermicide
    3. Intrauterine device (IUD)
    4. Tubal ligation
    5. Hormone-based contraceptive Note: For female participants receiving ritonavir or cobicistat, estrogen-based contraceptives are not reliable and an alternative method should be suggested.
21. Men and women not of reproductive potential are eligible without requiring the use of contraceptives. Acceptable documentation detailing sterilization and menopause are specified below.

    Note: Men who have sex with men only will not be required to use contraception. Note: Women who have sex with women only will not be required to use contraception.

    Note: Written/oral documentation communicated by clinician/clinician's staff of one of the following:
    1. Physician report/letter
    2. Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
    3. Discharge summary
    4. Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory
22. Agrees not to enroll on another study of an investigational agent during the study period, defined as any unlicensed investigational drug not yet approved for use in humans.
23. Willingness to defer routine vaccination, including influenza, from 14 days prior to enrollment through Day 56 of the study.

    Note: Individuals who require vaccination will delay enrollment until 14 after vaccination.
24. Agrees to refrain from blood donation during the course of the study.
25. Participants with Type 2 diabetes must have a hemaglobin A1C <8 within 12 months prior to screening.
26. Adequate organ function as indicated by the laboratory values provided in Table 16 of the protocol.

Exclusion Criteria:

1. Women of childbearing age/potential who are breast feeding, pregnant, or planning pregnancy from enrollment to 4 months after the last vaccination at D28, D196.
2. Untreated syphilis infection defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment. Note: Potential participants may rescreen with documentation of adequate treatment. Participants reporting symptoms consistent with syphilis infection between the screening visit and the vaccination visit should be assessed to determine the need for repeat testing prior to vaccination.
3. Current treatment for HCV or HCV treatment within 6 months prior to enrollment.
4. HIV RNA =150 copies/mL in the 6 months prior to screening.
5. Received any infusion blood product or hematopoetic growth factors within 6 months prior to enrollment.

   Note: receipt of COVID convalescent plasma >/= 90 days prior to screening is not enrollment is not exclusionary.
6. Use of any of the following agents within 90 days prior to enrollment: immunomodulatory, cytokine, or growth stimulating factors such as systemic cytotoxic chemotherapy or immune globulin.
7. Intent to use immunomodulatory treatment during the study.
8. Use of systemic corticosteroids or topical steroids over a total area exceeding 225 cm2 within 30 days prior to enrollment, or anticipated need for periodic use of systemic corticosteroids during the study.

   Note: Participants receiving stable physiologic doses of glucocorticoids, defined as the equivalent of prednisone =10 mg/day, will not be excluded. Participants receiving inhaled, intranasal, topical (as defined), intermittent intra-articular corticosteroids, or topical imiquimod will not be excluded.

   Note: Concomitant use of oral/systemic /intra-articular/inhaled/intranasal corticosteroids is prohibited for participants receiving ritonavir or cobicistat.
9. Use of any investigational HIV vaccine or HIV immunotherapy. Note: Exceptions allowed per PI review and approval.
10. Any experimental non-HIV vaccination within the 6 months prior to enrollment. Note: receipt of FDA or Emergency Use Authorization (EUA) approved or licensed COVID-19 vaccines is not exclusionary if = 14 days prior to enrollment on a case by case review by PI or designee.
11. Prior receipt of any adenovirus Group E-vectored vaccines including those for COVID-19 (i.e. AZD1222/AstraZeneca).

    Note: Prior immunization with smallpox vaccine is not exclusionary. Note: Janssen Ad26COVS1 COVID-19 vaccine is not exclusionary.
12. Prior receipt of a live attenuated vaccine received within 60 days prior to screening (i.e.varicella, measles, mumps, rubella (MMR), and yellow fever).

    Note: Individuals who require live vaccination will delay screening until 60 days after vaccination.

    Note: Receipt of Mpox vaccine is not exclusionary as long as the last Mpox vaccination is received at least 60 days prior to enrollment.
13. Use of any other investigational treatment within 6 months prior to enrollment, with the exception of Phase II or higher studies of antiretroviral agents.

    Note: Co-enrollment with other studies under an IND using an FDA approved medication that are not otherwise listed as prohibited will be considered on a case-by-case basis.
14. For any serious illness requiring systemic treatment or hospitalization, the participant must either complete therapy or be clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to enrollment.
15. History of inflammatory diseases involving the peripheral or central nervous system, including but not limited to Guillain-Barré Syndrome (GBS), myasthenia gravis, optic neuritis, multiple sclerosis, transverse myelitis, neuromyelitis optica spectrum disorder (NMOSD) and chronic inflammatory demyelinating polyneuropathy (CIDP), that in the opinion of the investigator would preclude participation.
16. History of pregnancy, head trauma or major surgery within 90 days prior to enrollment, that in the opinion of the investigator would preclude participation.

    Note: Minor surgery within 90 days prior to screening and not resulting in reduced mobility will be assessed on a case-by-case basis.
17. Any clinically significant acute or chronic medical condition, other than HIV infection, that in the opinion of the investigator would preclude participation.
18. History of malignancy within the last 3 years. Note: History of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary with documentation of resolution per topical treatment or complete resection as determined by a dermatologist at least 3 months prior to enrollment.
19. Immune deficiency other than that caused by HIV infection.
20. Any medical, psychiatric, substance abuse, occupational or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or assessment of safety.
21. Blood pressure consistently > 150 mm Hg systolic and >100 mm Hg diastolic. Note: Elevated BP during leukapheresis procedures is not exclusionary. Isolated elevations must be noted as acceptable and signed by study PI or designee.
22. History of seizure(s) within the past 3 years.
23. History of splenectomy.
24. Bleeding disorder including factor deficiency, coagulopathy or platelet disorder that requires special precautions (easy bruising without a formal diagnosis is not exclusionary) or on chronic anticoagulation.
25. Allergy to eggs and/or egg products.
26. History of anaphylaxis or severe adverse reaction to prior vaccines including symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
27. History of hereditary angioedema, acquired angioedema or idiopathic angioedema.
28. Known allergy/sensitivity or hypersensitivity to components of study vaccines.
29. Unstable asthma (e.g. sudden acute attacks occurring without an obvious trigger) or asthma requiring:

    1. Daily steroid or long-acting beta-agonist prevention
    2. Hospitalization in the last two years
30. Active chronic skin problems such as eczema or psoriasis not controlled with topical treatments.
31. Inability to communicate effectively with study personnel.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Gay, MD, MPH, Principal Investigator — University of North Carolina; Nilu Goonetilleke, PhD, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina at Chapel Hill (UNC).
Supporting Information: ICF
Time Frame: 9-36 months after publication
Access Criteria: Noted above
URL: http://unc.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Started | 8 | 8 | 2
Enrollment Leukapheresis | 8 | 8 | 2
Day 0 Vaccination | 8 | 8 | 2
Day 28 Vaccination | 8 | 8 | 2
Day 56 Leukapheresis/Large Volume Blood Draw | 8 | 8 | 2
Completed | 8 | 8 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes participants that were randomized to one of three study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 2 | 18
Age, Continuous [Median (Full Range); unit: years] | 58 [45 to 62] | 33.5 [24 to 67] | 50.5 [49 to 52] | 50 [24 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 6 | 8 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 2 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 2 | 8
  White | 4 | 6 | 0 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Grade 3 or Higher Treatment-Related Adverse Event (AE)
Description: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 was used to measure safety where Grade 1 is defined as mild, Grade 2 is defined as moderate, Grade 3 is defined as severe, and Grade 4 is defined as potentially life-threatening. Treatment-Related AEs were assessments that were considered related to study product as possible, probable, or definite as defined in the protocol. Confidence intervals around percentages were estimated using the Clopper-Pearson exact method.
Time Frame: First day of study treatment through 28 days following last vaccination, an average of 2 months
Population: All participants that received C62-M4, C1C62-M3M4, or placebo were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- C62-M4: C62 vaccine administered at Day 0, followed by M4 vaccine administered at Day 28
- C1C62-M3M4: C1 and C62 vaccines administered at Day 0, followed by M3 and M4 vaccines administered at Day 28
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 8 | 8 | 2
percentage of participants | 12.5 [0.32 to 52.7] | 0 [0 to 36.9] | 0 [0 to 84.2]

2. Secondary Outcome: Percent of Participants With a Grade 1 or Higher Treatment-Related Adverse Event (AE)
Description: as for outcome 1
Time Frame: First day of study treatment through day 196 (20 weeks following second vaccination), an average of 7 months
Population: All participants that received C62-M4, C1C62-M3M4, or placebo were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 8 | 8 | 2
percentage of participants | 87.5 [47.4 to 99.7] | 100 [63.1 to 100] | 50 [1.3 to 98.7]

3. Secondary Outcome: Median Fold-change in Magnitude of T-cell Response to HIV-1 Mosaic-1 Immunogen
Description: Relative changes in magnitude of T-cell responses to HIV-1 conserved region (Mosaic-1) between baseline (one or more of screening, enrolment, pre-vaccination leukapheresis or day 0) and day 35 was measured by ex vivo interferon (IFN)-gamma ELISpot. The relative change within participants (per vaccinated arm) was estimated using a geometric mean ratio and evaluated using either a Wilcoxon signed rank test (within-arm) or Wilcoxon rank-sum test (between-arm).
Time Frame: Baseline to day 35
Population: Participants who received C62-M4 or C1C62-M3M4 vaccines were included. Placebo participants' samples were collected to maintain blinding but excluded per the analysis plan, as the study focused on (i) changes from baseline to post-vaccination and (ii) differences between vaccine groups.
Measure: Median (Inter-Quartile Range); unit: log2 fold change
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 8 | 8 | 0
log2 fold change | 1.15 [0.32 to 1.92] | 1.66 [1.29 to 2.26] |
Statistical Analysis 1: Comparison: C62-M4 vs C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-1 from baseline to day 35 within all vaccinees is zero; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Within-group log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.63, 95% CI 2-sided [0.67 to 2.14]
Statistical Analysis 2: Comparison: C62-M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-1 from baseline to day 35 within the C62-M4 vaccinated arm is zero; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; median log2 fold change = 1.15, 95% CI 2-sided [0.09 to 2.59]
Statistical Analysis 3: Comparison: C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-1 from baseline to day 35 within the C1C62-M3M4 vaccinated arm is zero; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Within-am log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.66, 95% CI 2-sided [0.93 to 4.59]
Statistical Analysis 4: Comparison: C62-M4 vs C1C62-M3M4; The contrast is the magnitude of the T-cell response to Mosaic-1 from baseline to day 35 in C62-M4 versus C1C62-M3M4.The null hypothesis is that he distributions of the T-cell response to Mosaic-1 from pre-vaccination to day 35 are the same between the two vaccinated arms; Test type: Superiority; p = 0.279, Wilcoxon (Mann-Whitney); Between-arm comparisons in log2 fold changes were statistically assessed using a two-sided exact Wilcoxon rank-sum test

4. Secondary Outcome: Median Fold-change in Magnitude of T-cell Response to HIV-1 Mosaic-2 Immunogen
Description: Relative changes in magnitude of T-cell responses to HIV-1 conserved region (Mosaic-2) between baseline (one or more of screening, enrolment, pre-vaccination leukapheresis or day 0) and day 35 was measured by ex vivo IFN-gamma ELISpot. The relative change within participants (per vaccinated arm) was estimated using a geometric mean ratio and evaluated using either a Wilcoxon signed rank test (within-arm) or Wilcoxon rank-sum test (between-arm).
Time Frame: Baseline to day 35
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log2 fold change
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 8 | 8 | 0
log2 fold change | 1.79 [1.06 to 1.92] | 1.66 [1.16 to 2.26] |
Statistical Analysis 1: Comparison: C62-M4 vs C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-2 from baseline to day 35 within all vaccinees is zero; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Within-group log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.66, 95% CI 2-sided [1.09 to 2.33]
Statistical Analysis 2: Comparison: C62-M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-2 from baseline to day 35 within the C62-M4 vaccinated arm is zero; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.79, 95% CI 2-sided [0.59 to 3.40]
Statistical Analysis 3: Comparison: C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-2 from baseline to day 35 within the C1C62-M3M4 vaccinated arm is zero; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.66, 95% CI 2-sided [0.94 to 3.09]
Statistical Analysis 4: Comparison: C62-M4 vs C1C62-M3M4; The contrast is the magnitude of the T-cell response to Mosaic-2 from baseline to day 35 in C62-M4 versus C1C62-M3M4.The null hypothesis is that he distributions of the T-cell response to Mosaic-2 from pre-vaccination to day 35 are the same between the two vaccinated arms; Test type: Superiority; p = 0.878, Wilcoxon (Mann-Whitney); Between-arm comparisons in log2 fold changes were statistically assessed using a two-sided exact Wilcoxon rank-sum test

5. Secondary Outcome: Median Fold-change in Magnitude of T-cell Response to HIV-1 Mosaic-1 Immunogen
Description: Relative changes in magnitude of T-cell responses to HIV-1 conserved region (Mosaic-1) between baseline (one or more of screening, enrolment, pre-vaccination leukapheresis or day 0) and day 42 was measured by ex vivo IFN-gamma ELISpot. The relative change within participants (per vaccinated arm) was estimated using a geometric mean ratio and evaluated using either a Wilcoxon signed rank test (within-arm) or Wilcoxon rank-sum test (between-arm).
Time Frame: Baseline to day 42
Population: Participants who received C62-M4 or C1C62-M3M4 vaccines were included. One participant in the C1C62-M3M4 arm missed the collection visit at day 42 and was unevaluable for this outcome. Placebo participants' samples were collected to maintain blinding but excluded per the analysis plan, as the study focused on (i) changes from baseline to post-vaccination and (ii) differences between vaccine groups.
Measure: Median (Inter-Quartile Range); unit: log2 fold change
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 8 | 7 | 0
log2 fold change | 1.09 [0.50 to 1.89] | 2.00 [1.03 to 3.47] |
Statistical Analysis 1: Comparison: C62-M4 vs C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-1 from baseline to day 42 within all vaccinees is zero; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Within-group log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.47, 95% CI 2-sided [0.54 to 2.63]
Statistical Analysis 2: Comparison: C62-M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-1 from baseline to day 42 within the C62-M4 vaccinated arm is zero; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.09, 95% CI 2-sided [0.39 to 3.61]
Statistical Analysis 3: Comparison: C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-1 from baseline to day 42 within the C1C62-M3M4 vaccinated arm is zero; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 2.00, 95% CI 2-sided [0.43 to 4.37]
Statistical Analysis 4: Comparison: C62-M4 vs C1C62-M3M4; The contrast is the magnitude of the T-cell response to Mosaic-1 from baseline to day 42 in C62-M4 versus C1C62-M3M4.The null hypothesis is that he distributions of the T-cell response to Mosaic-1 from pre-vaccination to day 42 are the same between the two vaccinated arms; Test type: Superiority; p = 0.189, Wilcoxon (Mann-Whitney); Between-arm comparisons in log2 fold changes were statistically assessed using a two-sided exact Wilcoxon rank-sum test

6. Secondary Outcome: Median Fold-change in Magnitude of T-cell Response to HIV-1 Mosaic-2 Immunogen
Description: Relative changes in magnitude of T-cell responses to HIV-1 conserved region (Mosaic-2) between baseline (one or more of screening, enrolment, pre-vaccination leukapheresis or day 0) and day 42 was measured by ex vivo IFN-gamma ELISpot. The relative change within participants (per vaccinated arm) was estimated using a geometric mean ratio and evaluated using either a Wilcoxon signed rank test (within-arm) or Wilcoxon rank-sum test (between-arm).
Time Frame: Baseline to day 42
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: log2 fold change
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 8 | 7 | 0
log2 fold change | 1.57 [1.06 to 1.89] | 1.78 [0.96 to 3.47] |
Statistical Analysis 1: Comparison: C62-M4 vs C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-2 from baseline to day 42 within all vaccinees is zero; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Within-group log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.78, 95% CI 2-sided [0.81 to 2.51]
Statistical Analysis 2: Comparison: C62-M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-2 from baseline to day 42 within the C62-M4 vaccinated arm is zero; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.57, 95% CI 2-sided [0.63 to 3.89]
Statistical Analysis 3: Comparison: C1C62-M3M4; The null hypothesis is that the median log2-fold change in magnitude of T-cell response to Mosaic-2 from baseline to day 42 within the C162-M3M4 vaccinated arm is zero; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney); Within-arm log2 fold changes were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median log2 fold change = 1.78, 95% CI 2-sided [0.70 to 3.79]
Statistical Analysis 4: Comparison: C62-M4 vs C1C62-M3M4; The contrast is the magnitude of the T-cell response to Mosaic-2 from baseline to day 42 in C62-M4 versus C1C62-M3M4.The null hypothesis is that he distributions of the T-cell response to Mosaic-2 from pre-vaccination to day 42 are the same between the two vaccinated arms; Test type: Superiority; p = 0.955, Wilcoxon (Mann-Whitney); Between-arm comparisons in log2 fold changes were statistically assessed using a two-sided exact Wilcoxon rank-sum test

7. Secondary Outcome: Median Change in Breadth of T-cell Responses Targeting Conserved HIV-1 Immunogen Subpools
Description: Change in breadth of T-cell response was measured as the difference in the number of ex vivo reactive subpools (P076, PP077, PP078, PP079, PP080) from baseline (one or more of screening, enrolment, pre-vaccination leukapheresis or day 0) to post-vaccination (day 56). The difference in reactive subpools within participants (per vaccinated arm) was estimated and the median value was evaluated using a Wilcoxon signed rank test (within-arm) or Wilcoxon rank-sum test (between-arm).
Time Frame: Baseline to day 56
Population: Participants that received the C62-M4 or C1C62-M3M4 vaccines were included. However, sufficient sample volume at day 56 was available for 2 participants in the C62-M4 arm and 4 participants in the C1C62-M3M4 arm; only the pooled analysis across C62-M4/C1C62-M3M4 was reported. Placebo participants' samples were collected to maintain blinding but excluded per the analysis plan, as the study focused on (i) changes from baseline to post-vaccination and (ii) differences between vaccine groups.
Measure: Median (Inter-Quartile Range); unit: subpools
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
Number analyzed (Participants) | 2 | 4 | 0
subpools | 1.0 [0.5 to 1.5] | 2.0 [1.25 to 2.5] |
Statistical Analysis 1: Comparison: C62-M4 vs C1C62-M3M4; The null hypothesis is that the median change in breadth of T-cell response to HIV-1 subpools from baseline to day 56 within all vaccinees is zero; Test type: Superiority; p = 0.125, Wilcoxon (Mann-Whitney); Within-group changes in breadth from baseline to day 56 were statistically assessed using a two-sided exact Wilcoxon signed rank test; Median Difference (Net) = 2, 95% CI 2-sided [-1 to 4]

ADVERSE EVENTS:
Time Frame: From time participants received the study intervention through Day 196.
Arm/Group | C62-M4 | C1C62-M3M4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C62-M4 (N=8) | C1C62-M3M4 (N=8) | Placebo (N=2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 4 (4) | 0 (0)
Fatigue (General disorders) | 6 (11) | 6 (12) | 1 (1)
Injection site erythema (General disorders) | 2 (4) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (3) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 5 (27) | 8 (50) | 1 (1)
Injection site swelling (General disorders) | 2 (4) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (2) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 2 (4) | 0 (0)
Malaise (General disorders) | 2 (4) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood HIV RNA increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 2 (4) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 7 (9) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT05604209/Prot_001.pdf
  • Statistical Analysis Plan (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT05604209/SAP_002.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT05604209/ICF_000.pdf